CLINICAL TRIAL: NCT00663741
Title: Phase I Study to Investigate Safety, Pharmacokinetics and Preliminary Efficacy Profile of Sorafenib (BAY 43-9006) in Combination With S-1 Plus CDDP in Asian Patients With Unresectable / Recurrent Gastric Cancer
Brief Title: Sorafenib Gastric Cancer Asian Phase I Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Head Clinical Pharmacology, Bayer Yakuhin, Ltd.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12931
Record Dates: First submitted 2008-04-17; First posted 2008-04-22 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Gastric Cancer
Keywords: Unresectable / recurrent gastric cancer; Sorafenib; S-1; Gastric; Cisplatin; CDDP
MeSH Terms: conditions — Stomach Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)
- Arm 2 (Experimental)
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)
- Arm 3 (Experimental)
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — Sorafenib (400 mg bid) + S-1 (40 mg/m2 bid, 3 weeks on / 2 weeks off) + CDDP (60 mg/m2 on Day 8) / 35 days / cycle
  Arms: Arm 1
Drug: Sorafenib (Nexavar, BAY43-9006) — Sorafenib (400 mg bid) + S-1 (25 mg/m2 bid, 3weeks on / 1 week off) + CDDP (75 mg/m2 on Day 1) / 28 days / cycle
  Arms: Arm 2
Drug: Sorafenib (Nexavar, BAY43-9006) — Sorafenib (400 mg bid) + S-1 (40 mg/m2 bid, 3 weeks on / 1 week off) + CDDP (75 mg/m2 on Day 1) / 28 days cycle
  Arms: Arm 3

SUMMARY:
This study is to investigate safety, pharmacokinetics and preliminary efficacy profile of sorafenib in combination with S-1 plus cisplatin in Asian patients with unresectable / recurrent gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmation of the primary unresectable or recurrent gastric cancer (both with and without measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) are allowed). Peritoneal dissemination without ascites is allowed.
* No prior systemic anticancer therapy including chemotherapy, immunotherapy, targeted agents or experimental therapies for advanced disease
* Prior adjuvant therapy/neo adjuvant therapy is allowed if recurrence occurred 6 months after completion of these therapies
* Age >/= 18 years and < 75 years

Exclusion Criteria:

* Known brain metastasis, spinal cord compression or meningeal carcinomatosis.
* Clinically relevant ascites
* Concurrent cancer that is distinct in primary site or histology from gastric cancer
* Any condition that impairs patient's ability to swallow whole pills

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-05; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Safety and pharmacokinetics | 20 weeks after start of treatment

SECONDARY OUTCOMES:
1 year survival rate | 1 year after start of treatment
Overall survival | 1 year after start of treatment
Progression free survival | 1 year after start of treatment
Response rate | 1 year after start of treatment
Duration of response | Time from initial Response to documented Tumor Progression

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (3):
- Japan (3):
  - Kashiwa, Chiba
  - Kobe, Hyōgo
  - Chuo-ku, Tokyo